CLINICAL TRIAL: NCT02004067
Title: Safety Study of the Use of Topical Cyclosporine in the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Rossen Mihaylov Hazarbassanov, MD, PhD, Researcher, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17821013.0.0000.5505
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Primary Sjogren Syndrome; Secondary Sjogren Syndrome; Aqueous Deficient Dry Eye Disease; Evaporative Dry Eye Disease
Keywords: Evaporative; Aqueous deficient; Dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins; Castor Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Refresh Endura (Active Comparator): Topical lubricant containing (glycerin; polysorbate 80; castor oil; carbomer, boric acid, sodium hydroxide, purified water), one drop 2 times a day, for 3 months.
  Interventions: Drug: Refresh Endura
- Restasis (Experimental): Topical immunomodulatory lubricant (Ophthalmic emulsion containing cyclosporine 0.5 mg/mL, i.e., 0.05%), one drop 2 times a day, for 3 months
  Interventions: Drug: Restasis

INTERVENTIONS:
Drug: Restasis — Restasis is an ophthalmic emulsion containing cyclosporine 0.5 mg/mL, produced by Allergan Inc.
  Other Names: Cyclosporine 0.05%
  Arms: Restasis
Drug: Refresh Endura — Refresh Endura is a topical lubricant produced by Allergan, Inc.
  Other Names: Castor oil
  Arms: Refresh Endura

SUMMARY:
In the present study the investigators aim to determine the efficacy of an immunomodulating topical medication, compared with a topical lubricant, on the treatment of dry eye disease (DED) due to primary or secondary Sjögren's syndrome (aqueous deficient DED) and evaporative DED.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and inflammation of the ocular surface. DED prevalence is estimated around 15 -35% of the population over 50 years old. There is a wide variety of topic medications for the treatment of DED, though few aim the re-establishment of tear osmolarity equilibrium and reduction of damages to the ocular surface. The treatment of DED can include a medical treatment, such as tear substitution, tear preservation, production stimulation, anti-inflammatory; it can also include surgical treatment, as tarsorrhaphy and salivary gland transplant. Considering tear substitutes and anti-inflammatory topical treatments, the purpose of our study is to determine efficacy of an immunomodulating topical medication containing 0.05% cyclosporine A (CsA), compared to a topical lubricant (vitamin A, Refresh Endura®), on the treatment of dry eye disease (DED) due to primary or secondary Sjögren's syndrome (aqueous deficient DED) and evaporative DED.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed for mild to moderate Aqueous Deficient DED (ADDED), defined as Schirmer 1 < 10mm;
* Patients diagnosed for mild to moderate Evaporative DED (EDED), defined as normal Schirmer 1 and BUT < 5 seconds;
* Patients submitted to refractive surgery,
* Patients capable of understanding instructions, signing the term of consent and available to attend all exam visits.

Exclusion Criteria:

* patients with punctual occlusion,
* active ocular infection or inflammatory disease,
* history of herpetic keratitis,
* contact lens use during trial period,
* patients with glaucoma,
* any eyelid globe malposition abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Ocular surface inflammation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rossen M Hazarbassanov, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Departamento de Oftalmologia da Escola Paulista de Medicina - UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided